CLINICAL TRIAL: NCT03439566
Title: Does Preoperative Pain Levels by Venipuncture Predict Late Postoperative Pain Levels? - a Prospective Cohort Study of Total Hip Arthroplasty Patients at Zealand University Hospital, Koege
Brief Title: Does Preoperative Pain Levels by Venipuncture Predict Late Postoperative Pain Levels?
Status: Completed | Type: Observational
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Anja Geisler, PhD student/ clinical nurse specialist, Zealand University Hospital
Other Study IDs: SM4-AG-17
Record Dates: First submitted 2017-11-24; First posted 2018-02-20 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Pain, Postoperative
Keywords: pain measures; prediction of pain; pain management
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Total hip arthroplasty: No intervention will take place. Only registration and data collection of patient´s care and treatment will take place. There will be no changes in patient´s treatment.

SUMMARY:
This study wishes to investigate if pain by peripheral venous cannulation (PVC) preoperatively, will predict pain levels after 24 h postoperatively. Furthermore, to investigate moderate/severe pain at the postoperatively at the post-anaesthesia care unit (PACU) is associated with increased late (24h) pain. Additionally, if the PACU nurse is able to predict if the patient will be a high pain responder, by using a clinical judgement. Finally to evaluate the patient's pain-levels at home after discharge and investigate for associations between postoperative pain and post-discharge pain.

DETAILED DESCRIPTION:
Postoperative pain remains insufficiently treated in clinically relevant proportions of patients across procedures, but with varying incidences. Preoperative identification of patients at risk for increased postoperative pain may result in stratification of perioperative analgesic protocols, aiming at reducing pain in high-risk patients while avoiding over-treatment in those at low-risk.

Several potential patient-related factors have been suggested as associated with an increased risk of higher postoperative pain levels. Studies indicate a positive correlation between postoperative pain levels and e.g. preoperative pain levels, gender, age and socioeconomically and psychological variables. The Pain Catastrophizing Scale (PCS), has been used to look for associations between psychological variables and levels of early and late pain as well. However, no firm data exist for a clinically useful identification of individual high pain responders.

Preoperative sensory testing of patient's nociception has the potential to predict postoperative pain levels. However, a review dealing with the prediction of postoperative pain based on experimental pain studies demonstrated that quantitative sensory testing was only able to predict 4 - 54% of the variance of the postoperative pain of individual patients. Another recent study of clinically applicable tests suggested that relevant sensitivity and specificity can be achieved, but this has not been translated into clinical practice or confirmed. Thus, no preoperative testing method has proven clinically relevant or useful until now.

A newer pragmatic clinical study indicated that the pain intensity associated with peripheral venous cannulation (PVC) could be used as a simple predictor of the magnitude of early pain levels at one hour postoperatively at the post-anaesthesia care unit (PACU). That study, however, did not test the possible association between venepuncture related pain and later pain levels at 24h.

Another simple method for early identification of those with an intensified need of pain treatment after PACU discharge could be to investigate if higher pain levels early postoperatively at the PACU are associated with higher levels of late postoperative pain. Especially, we find it relevant at the individual patient level to investigate if NRS below 3 (moderate/severe pain) in the early postoperative phase at the PACU is associated with NRS levels above 3 late postoperatively.

Also, it could be relevant to investigate if the PACU-nurses, based on their clinical evaluation, are able to predict if the patient would experience an increased risk of moderate/severe pain after PACU discharge. Such a simple clinical tool of staff's judgement of risk of postoperative pain levels has never been tested before.

The hypothesis is that levels of early and late pain are associated and with a simple clinical related tool it could be possible to identify patients with increased pain levels at 24-hours postoperatively.

With updated fast-track perioperative patient causes, patients often are discharged quickly after the surgical procedure. Often there may be a lack of knowledge on how they manage to return to daily living. Pain can be a major problem for the patients, possibly also at home.

Even though one cannot be certain that patients with severe pain, will contact the hospital after discharge. Not only can pain delay rehabilitation it can also be a major factor for developing chronic pain.

Therefore, it is relevant to monitor the patient's pain-levels, quality of sleep, mood, as well as analgesic use and side-effects at home, using a diary from discharge until 5 days postoperatively. Especially, to investigate if patients with higher postoperative pain levels also experience excess pain-related problems after discharge.

.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing total hip arthroplasty in spinal anaesthesia
* Patients who understand and speak Danish or English

Exclusion Criteria:

* Patients who cannot cooperate with the study
* Alcohol and drug dependency as judged by the investigator
* Patients in need of urgent surgery
* Patients whom first Peripheral Venous Cannulation attempt was unsuccessful

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing total hip arthroplasty (THA) at Zealand University Hospital, Koege meeting the inclusion criteria
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Difference between groups, in levels of pain (NRS < / > 2) by peripheral venous cannulation (PVC) preoperatively, during mobilisation at 24 hour postoperatively | Preoperatively just before the patient will be sedated and 24h postoperatively
  The patients will be divided in two groups when the peripheral venous cannula is placed Group 1 is patients with a NRS pain below 2. Group 2 is patients with NRS levels above 2. Is there a correlation between the groups when looking at the NRS levels at rest after the spinal has ceased and at 24h mobilisation postoperatively

SECONDARY OUTCOMES:
Difference between groups, defined by levels of pain by peripheral venous cannulation (PVC) preoperatively (NRS < / > 2) at rest, after spinal has ceased (Bromage=0-1), at 24 h postoperatively | Preoperatively, just before the patient will be sedated when the spinal has ceased (Bromage=0-1) at 1 to 4 h postoperatively and at 24h postoperatively
  The patients will be divided in two groups when the PVC is placed according to NRS level Is there a correlation between the groups when looking at the NRS levels at rest after the spinal has ceased and at 24h postoperatively and opioid consumption?
Difference between groups, defined by Post Anaesthesia Care Unit nurses´ prediction of high pain responders (yes/ no), and levels of pain at 24-hour postoperatively, at rest and during mobilisation, and 24h postoperative opioid consumption | Postoperatively at discharge from the PACU up to 4h postoperatively and 24 hours postoperatively
  The patients will be divided in two groups when the peripheral venous cannula is placed. Group 1 is patients with a NRS pain below 2. Group 2 is patients with NRS levels above 2. Is there a correlation between the groups and the PACU nurse´s prediction about the patient beeing a high pain responder or not and NRS levels of pain at rest and during mobilisation at 24 h postoperatively and 24 h opioid consumption.
Difference between groups, defined by patient's experienced level of pain at rest (Numerical ranking scale < 3 / > 3) and levels of pain at rest at 24 hour postoperatively and 24-hour postoperative opioid consumption. | 24 hour postoperatively
  The patients will be divided in two groups patients with NRS pain levels below 3 and above 3. Is there a correlation between the groups when looking at the NRS levels at rest at 24h postoperatively and 24 h opioid consumption?
A patient diary, investigating postoperative pain levels, sleep and mood | Day 1 to 5 postoperatively
  Pain monitored using NRS. Nausea monitored using Verbal Rating Scale (None, slightly, moderate, severe) Vomiting monitored by numbers of. Medication monitored in mg. Patients mood monitored by yes or no. Quality of sleep monitored by good sleep, difficulties sleeping, many awakenings, no sleep at all

CONTACTS AND LOCATIONS:
Overall Officials: Anja Geisler, PhD student, Principal Investigator — Zealand University Hospital, Koege
Locations (1):
- Zealand University Hospital, Koege, Copenhagen, Køge, Denmark

REFERENCES:
- [Derived] Geisler A, Zachodnik J, Laigaard J, Kruuse LS, Sorensen CV, Sandberg M, Persson EI, Mathiesen O. Using four different clinical tools as predictors for pain after total hip arthroplasty: a prospective cohort study. BMC Anesthesiol. 2020 Mar 3;20(1):57. doi: 10.1186/s12871-020-00959-2. PMID 32126971